CLINICAL TRIAL: NCT02511730
Title: A Multi-Reader Multi-Case Controlled Clinical Trial to Evaluate the Comparative Accuracy of the Fujifilm Full Field Digital Mammography (FFDM) Plus Digital Breast Tomosynthesis (DBT) Versus FFDM Alone in the Detection of Breast Cancer
Brief Title: Pilot Mammography Reader Study to Assess Breast Cancer Detection in FFDM Plus DBT Versus FFDM Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujifilm Medical Systems USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: FMSU2013-004E
Record Dates: First submitted 2015-07-23; First posted 2015-07-30 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: Mammography
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FFDM Plus DBT (Experimental): Breast Images with FFDM and DBT
  Interventions: Device: FFDM Plus DBT
- FFDM Alone (Active Comparator): Breast Images with FFDM alone
  Interventions: Device: FFDM

INTERVENTIONS:
Device: FFDM Plus DBT — FujiFilm Aspire Cristalle System
  Arms: FFDM Plus DBT
Device: FFDM — FujiFilm Aspire Cristalle System
  Arms: FFDM Alone

SUMMARY:
The purpose of this pilot is to provide credible performance estimate information in order to conduct subsequent reader studies.

DETAILED DESCRIPTION:
This pilot reader study was to determine the following:

1. the radiologist's performance metrics for the two reading modalities, i.e., "FFDM read on the Aspire Bellus workstation" and "FFDM read in conjunction with DBT read on the Aspire Bellus workstation",;
2. the magnitude and direction of differences between performance metrics for the two modalities; and
3. variance components and correlations that would influence samples sizes and case mix for the subsequent pivotal reader study comparing performance metrics between the two modalities.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects participating in FMSU004A protocol with known clinical status

Exclusion Criteria:

* Subjects with unknown clinical status not participating in FMSU004A protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Uzenoff, Study Director — Fujifilm Medical Systems USA, Inc.
Locations (4):
- United States (4):
  - Scottsdale Medical Imaging, Limited (SMIL), Scottsdale, Arizona
  - Elizabeth Wende Breast Care, LLC (EWBC), Rochester, New York
  - University of North Carolina - at Chapel Hill, Chapel Hill, North Carolina
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The 100 breast screening and diagnostic cases selected for this study, were obtained from the FMSU2013-004A acquisition study. The statistician randomly selected cases to provide a distribution of density, finding types, etc.
Pre-assignment Details: Each radiologist read all 100 cases as FFDM only and FFDM+DBT(100 cases multiplied by 2 modalities = 200 reads) with a 4 week washout period between the 2 sessions.
Groups:
- FFDM Plus DBT, Then FFDM Only: Readers to read half of the FFDM plus DBT images followed by half of the FFDM only images at each of the 2 sessions. There was a 4 week memory washout period between the 2 sessions.
- FFDM Only, Then FFDM Plus DBT: Readers to read half of the FFDM only images followed by half of the FFDM plus DBT images at each of the 2 sessions. There was a 4 week memory washout period between the 2 sessions.
Period: First Reading Session
Arm/Group | FFDM Plus DBT, Then FFDM Only | FFDM Only, Then FFDM Plus DBT
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: 4 Week Memory Washout Period
Arm/Group | FFDM Plus DBT, Then FFDM Only | FFDM Only, Then FFDM Plus DBT
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0
Period: Session Reading Session
Arm/Group | FFDM Plus DBT, Then FFDM Only | FFDM Only, Then FFDM Plus DBT
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 100 study participants (resulting in 200 images) in total who had their images reviewed by 6 radiologist readers. Images were acquired under acquisition study FMSU2013-004A.
Groups:
- All 100 Cases/Study Participants: Each case contributed 2 sets of images: FFDM only as well as DBT plus FFDM. Therefore there were 200 reads acquired from the 100 cases/participants.
Arm/Group | All 100 Cases/Study Participants
Number analyzed (Participants) | 100
Age, Customized [Mean (Standard Deviation); unit: years]
  Participant Age | 58 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3
  Black or African American | 8
  White | 87
  Other/Unknown | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Compare Per Subject Area Under Curve (AUC): FFDM Only vs DBT Plus FFDM
Description: Breast AUC performance metrics to determine if FFDM plus DBT improved cancer detection rate, requiring correct lesion localization. Statistician to estimate AUCs for each reader in each review condition (FFDM read in conjunction with FFDM plus DBT read) based on their Probability of Malignancy (POM) scores. POM scores will require correct lesion localization, such that in a case with cancer if the reader recorded one or more findings in the case but none of them are determined by the truther to match the location(s) of any proven malignancies, a POM score of 0 will be assigned to the case. Statistician to provide graphical representations of each reader's ROC curve for each review condition. For each reader the difference between the AUC for the FFDM read in conjunction with the FFDM plus DBT will be presented. Statistician to perform MRMC comparison of AUC's between FFDM read in conjunction with FFDM plus DBT using the MRMC method of Dorfman, Berbaum & Metz (1992).
Time Frame: 1 month
Population: The study employed a fully factorial, counterbalanced crossover design in which all readers reviewed images from all cases in two visits separated by a memory washout period of approximately 4 weeks. Each reader read half FFDM cases and half FFDM + DBT cases during each of 2 visits.
Measure: Mean (Standard Error); unit: Probability
Groups:
- FFDM: Breast Images with FFDM alone
  FFDM: Fujifilm Aspire Cristalle System
Arm/Group | FFDM Plus DBT | FFDM
Number analyzed (Participants) | 100 | 100
Probability | 100 (0.812) | 100 (0.780)

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: There were no AE's expected for this study, as it was a radiologist reader study utilizing retrospective imaging. No study subjects were on-site for this retrospective review. No Adverse Events to report.
Arm/Group | FFDM Plus DBT | FFDM
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No